CLINICAL TRIAL: NCT04438642
Title: Biological and Esthetic Evaluation of Ceramic Onlay With Different Preparation Designs (A Randomized Controlled Clinical Trial)
Brief Title: Biological and Esthetic Evaluation of Ceramic Onlay With Different Preparation Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ahmed Adel Mahmoud Gadallah (Other)
Responsible Party: Sponsor-Investigator, Ahmed Adel Mahmoud Gadallah, PhD researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gadallah
Record Dates: First submitted 2020-02-25; First posted 2020-06-19 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Unsatisfactory Restoration of Tooth; Carious Teeth
Keywords: ceramic onlay; conventional preparation; conservative preparation; Butt joint with bevel; shoulder finish line; biologic response
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional ceramic onlay with shoulder finishline (Other): tooth that need ceramic onlay restoration, a conventional cavity will be prepared with shoulder finishline.
  Interventions: Procedure: shoulder finishline
- conservative ceramic onlay preparation buttjoint with bevel (Experimental): tooth that need ceramic onlay restoration, a conservative cavity will be prepared with butt joint with bevel finishline.
  Interventions: Procedure: butt joint with bevel

INTERVENTIONS:
Procedure: shoulder finishline — tooth will be prepared having shoulder finishline.
  Arms: conventional ceramic onlay with shoulder finishline
Procedure: butt joint with bevel — tooth will be prepared having butt joint with bevel finishline.
  Arms: conservative ceramic onlay preparation buttjoint with bevel

SUMMARY:
Aim of study: is to asses biological and esthetical success of ceramic onlay restorations while preparing the teeth using shoulder finish line preparation versus butt joint with bevel preparation.

Methods:

Patients with need to posterior onlay restoration (premolars and molars) will be allocated into two groups either conventional (shoulder finish line) or conservative group (butt joint with bevel), after tooth preparation impression, restoration fabrication, try in, cementation and restoration will be evaluated two weeks post cementation then follow up will be held every two months for 1 year.

DETAILED DESCRIPTION:
* Research objective: The aim of this study is to asses biological and esthetical success of ceramic onlay restorations while preparing the teeth using shoulder finish line preparation versus butt joint with bevel preparation.
* Research Procedure:

  * Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs and primary impression (alginate impression*) for diagnostic cast construction.
  * Visit 2: Tooth preparation according to its group either shoulder, or butt joint with bevel preparation, secondary impression using addition silicone rubber base material two step two viscosities technique and temporary restoration.
  * Visit 3: evaluation of e-max press onlay ceramic restoration on the cast then evaluation intra-oral on the prepared tooth and permanent cementation of the final restoration using adhesive resin cement.
  * Visit 4: Every 2 months post operatively follow-up visit for one year.
  * PICOTS P: Population: Patients requiring posterior onlays. I: Intervention: butt joint finish line with bevel preparation for ceramic onlay.

C: comparator: shoulder finish line preparation for ceramic onlay.

O: Outcome:

Primary: Postoperative sensitivity Secondary: Marginal discoloration Tertiary: Secondary Caries T: Time: 1 year. S: Study design: Randomized controlled clinical trial.

* Research question For patients requiring posterior onlays, does the use of conservative preparation offer better biological response and esthetics when compared to conventional onlay preparation?
* Participant timeline:
* The patient will be treated in visits designated as follows:

  * Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs and primary impression (alginate impression) for diagnostic cast construction.
  * Visit 2: Tooth preparation according to its group either shoulder, or butt joint with bevel preparation, secondary impression using addition silicone rubber base material two step two viscosities technique and temporary restoration.
  * Visit 3: evaluation of e-max press onlay ceramic restoration on the cast then evaluation intra-oral on the prepared tooth and permanent cementation of the final restoration using adhesive resin cement.
  * Visit 4: Every 2 months post operatively follow-up visit for one year.
* Allocation

Randomization:

- Simple randomization will be done using computerized random number generator

Allocation:

* Sequence generation
* A dental colleague will allocate the participant patients into two groups with 1:1 allocation ratio by using computerized Sequence generation
* Blinding
* Double blinding (trial participants and outcome assessor)
* Two dental colleague assessors who are blinded about the aim of the study and participant's allocation will be responsible for assessing the outcomes of this study.

Data collection methods:

* Primary 1ry: Postoperative sensitivity will be assessed by asking patients according to modified USPHS criteria and given a score (Alpha, Bravo)
* Secondary 2ry outcome: Marginal discoloration will be assessed according to modified USPHS criteria and given a score (Alpha, Bravo B1, Bravo B2, Charlie).
* Tertiary 3ry outcome: Secondary Caries will be assessed by visual and given a score (Alpha, Bravo).

Plans to promote participant retention & complete follow-up:

* The main investigator will record telephone numbers and address of the patients included in the study. All patients will be given a phone call before the next appointment. Many efforts will be done to promote participant retention such as, sending SMS greetings in the feasts, any celebration and in his/ her birthday.
* Data management
* The main investigator will enter patient data electronically. Patient files are to be stored in Numerical order in a secured place.
* Statistical methods
* Qualitative data will be presented as frequencies and percentages. Chi-square test or Fisher's Exact test when applicable will be used for comparisons related to qualitative variables. Friedman's test will be used to study the changes by time within each group. Dunn's test will be used for pair-wise comparisons when Friedman's test is significant.
* The significance level will be set at P ≤ 0.05. Statistical analysis will be performed with IBM® SPSS® Statistics Version 20 for Windows (SPSS, Inc., an IBM Company).

D) Data monitoring

* Monitoring
* The main supervisor is responsible of data monitoring if harms arise, interim analysis will be done.
* Harms
* The main investigator will record, document and treat any adverse effect like pain or even failure.
* Expected risk to the human subjects:

  1. Possibility of restoration dislodgment (the patient should keep the restoration and contact the researcher as soon as possible as the restoration will be assessed for cementation or replacement).
  2. Possibility of restoration fracture (the patient should keep the fractured part and contact the researcher as soon as possible as a new restoration will be placed).
  3. In case failure of the onlay restoration the tooth will be assessed for the new required restorative modality.
* Consent
* Researcher will discuss the trial with all patients. Patients will then be able to have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1-From 18-70 years old, be able to read and sign the informed consent document.30 2- Have no active periodontal or pulpal diseases, have teeth with good restorations.

  3- Psychologically and physically able to withstand conventional dental procedures 4- Patients with teeth problems indicated for posterior onlay (molars or premolars).
  1. Decayed teeth
  2. Teeth restored with large filling restorations 5- Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient less than 18 or more than 70 years
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene, high caries risk and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Lack of opposing dentition in the area of interest. 8- the presence of a removable or fixed orthodontic appliance, signs of bruxism or clenching, the absence of more than one unit in the posterior region.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-11-09 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
postoperative sensitivity | 1 year follow up
  pain immediately after restoration cementation

SECONDARY OUTCOMES:
Marginal Discoloration | 1 year follow up
  Margins between tooth and restoration have discoloration. Measuring device: visual and probe (used according to USPHS instructions)
  Measuring unit: Alpha, Bravo B1, Bravo B2, Charlie (according to USPHS measuring units) as following:
  Alpha: no discoloration along the margin.
  Bravo B1: discoloration noted along the margin less than 50 percent of exposed margin.
  Bravo B2: discoloration noted along the margin greater than 50 percent of exposed margin.
  Charlie: discoloration penetrating along the margin.

OTHER OUTCOMES:
secondary carries | 1 year follow up
  carries that is developed due to restoration Measuring device: visual and probe (used according to USPHS instructions)
  Measuring unit: Alpha and Bravo (according to USPHS measuring units) as following:
  Alpha: carries absent along the margin.
  Bravo: carries present along the margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Faculty Of Dentistry Fixed Prosthodontics clinic, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
the outcome results